CLINICAL TRIAL: NCT02297139
Title: Continuing Treatment for Subjects Who Have Participated on a Prior Protocol Investigating Dasatinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CA180-597
Record Dates: First submitted 2014-11-19; First posted 2014-11-21 (Estimated); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Multiple Indications Cancer
MeSH Terms: interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dasatinib (Experimental): This is a continuation roll-over study for patients receiving benefit from prior dasatinib protocols. All subjects will receive dasatinib as per previous protocol
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib

SUMMARY:
The purpose of this study is to continue to provide dasatinib to patients that are currently participating in another dasatinib trial that is ending and for which there is no other option to provide dasatinib.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Participated in and completed a previous dasatinib protocol (including but not limited to CA180056, CA180363 or CA180227) and is deemed by the investigator to be deriving benefit from dasatinib as defined by the previous protocol
* Receiving dasatinib at the time of signature of informed consent
* Males and Females, ages 18 and older

Exclusion Criteria:

* All patients previously discontinued from a dasatinib study for any reason
* Any serious or uncontrolled medical disorder or active infection that would impair the ability of the subject to receive protocol therapy
* History of allergy to dasatinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-07-31 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (6):
- Local Institution, Besançon, France
- Poland (5):
  - Local Institution - 0006, Krakow, Lesser Poland Voivodeship
  - Local Institution, Chorzów
  - Local Institution, Lodz
  - Local Institution - 0003, Warsaw
  - Local Institution - 0002, Wroclaw

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/us/en/home.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Prostate Cancer: Continuing treatment for prostate cancer participants who have participated on prior protocol CA180-227 investigating dasatinib. Dasatinib tablet administered once a day by mouth.
- Chronic Phase - Chronic Myeloid Leukemia (CP-CML): Continuing treatment for CP- CML participants who have participated on prior protocols CA180-363 and CA180-056 investigating dasatinib. Dasatinib tablet administered once a day by mouth.
Period: Overall Study
Arm/Group | Prostate Cancer | Chronic Phase - Chronic Myeloid Leukemia (CP-CML)
Started | 1 | 16
Completed | 0 | 0
Not Completed | 1 | 16
Not completed — Disease progression | 0 | 1
Not completed — Study drug toxicity | 0 | 4
Not completed — Participant request to discontinue study treatment | 0 | 1
Not completed — Maximum clinical benefit | 1 | 0
Not completed — Administrative reason by sponsor | 0 | 2
Not completed — Other reasons | 0 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prostate Cancer | Chronic Phase - Chronic Myeloid Leukemia (CP-CML) | Total
Number analyzed (Participants) | 1 | 16 | 17
Age, Continuous [Median (Full Range); unit: Years] | 58 [58 to 58] | 64.5 [35 to 75] | 62 [35 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 8 | 8
  Male | 1 | 8 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 15 | 15
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 16 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received Dasatinib Treatment
Description: Number of participants who received dasatinib treatment for prostate cancer and chronic phase chronic myeloid leukemia who had also participated on prior protocols CA180-227, CA180-363 and CA180-056 investigating dasatinib. Dasatinib tablet administered once a day by mouth.
Time Frame: From first dose on this study (CA180-597) to last dose on this study (up to approximately 76 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Prostate Cancer | Chronic Phase - Chronic Myeloid Leukemia (CP-CML)
Number analyzed (Participants) | 1 | 16
Participants | 1 | 16

2. Primary Outcome: Duration of Treatment
Description: Duration of treatment for participants who received dasatinib treatment for prostate cancer and chronic phase chronic myeloid leukemia who had also participated on prior protocols CA180-227, CA180-363 and CA180-056 investigating dasatinib. Dasatinib tablet administered once a day by mouth.
Time Frame: From first dose on this study (CA180-597) to last dose on this study (up to approximately 76 months)
Population: All treated participants
Measure: Median (Full Range); unit: Months
Arm/Group | Prostate Cancer | Chronic Phase - Chronic Myeloid Leukemia (CP-CML)
Number analyzed (Participants) | 1 | 16
Months | 25.3 [25.3 to 25.3] | 55.9 [4.0 to 75.5]

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of Participants with Adverse Events (AEs). An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug.
Time Frame: From first dose on this study (CA180-597) to 30 days after last dose of study therapy (up to approximately 77 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Prostate Cancer | Chronic Phase - Chronic Myeloid Leukemia (CP-CML)
Number analyzed (Participants) | 1 | 16
Participants | 1 | 15

4. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Number of participants with serious adverse events (SAEs). SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: From first dose on this study (CA180-597) to 30 days after last dose of study therapy (up to approximately 77 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Prostate Cancer | Chronic Phase - Chronic Myeloid Leukemia (CP-CML)
Number analyzed (Participants) | 1 | 16
Participants | 0 | 8

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their first dose until their study completion (up to approximately 82 months). SAEs and other AEs were assessed from first dose to 30 days after last dose of study therapy (up to approximately 77 months).
Arm/Group | Prostate Cancer | Chronic Phase - Chronic Myeloid Leukemia (CP-CML)
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/16
Serious Adverse Events (participants affected / at risk) | 0/1 | 8/16
Other Adverse Events (participants affected / at risk) | 1/1 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prostate Cancer (N=1) | Chronic Phase - Chronic Myeloid Leukemia (CP-CML) (N=16)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Drug hypersensitivity (Immune system disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prostate Cancer (N=1) | Chronic Phase - Chronic Myeloid Leukemia (CP-CML) (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 2
Fatigue (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 3
COVID-19 (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 4
Urinary tract infection (Infections and infestations) | 0 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Blood testosterone increased (Investigations) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 1
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 6
Phlebitis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-19): https://cdn.clinicaltrials.gov/large-docs/39/NCT02297139/Prot_SAP_000.pdf